CLINICAL TRIAL: NCT06014021
Title: Treatment of Urinary Incontinence and Other Pelvic Floor Dysfunctions in Female Athletes
Brief Title: Tele-rehabilitation for Female Athletes With Pelvic Floor Dysfunctions
Acronym: ACTITUD2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Collaborators: Fundació d'investigació Sanitària de les Illes Balears (Other Government); Consejo Superior de Deportes, Spain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 124CER19_
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Pelvic Floor Disorders
Keywords: Female; Athletes; Track and Field; Tele-rehabilitation; Strengthening
MeSH Terms: conditions — Pelvic Floor Disorders | interventions — Health Personnel

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The design of this study does not allow to mask participants or care providers. Investigators or outcomes assessors will not know which group athletes belong.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 (Experimental): All participants will use an Smartphone application with access to information about pelvic floor and communication with healthcare team, and a strengthening program for PF, while using an intracavitary biofeedback device.
  Interventions: Behavioral: Pelvic floor muscle training with biofeedback device; Behavioral: Information about pelvic floor and communication with health professionals
- Experimental group 2 (Active Comparator): All participants will use an Smartphone application with access to information about pelvic floor and communication with healthcare team, and a strengthening program for PF.
  Interventions: Behavioral: Pelvic floor muscle training; Behavioral: Information about pelvic floor and communication with health professionals
- Control group (Active Comparator): All participants will use an Smartphone application with access to information about pelvic floor and communication with healthcare team.
  Interventions: Behavioral: Information about pelvic floor and communication with health professionals

INTERVENTIONS:
Behavioral: Pelvic floor muscle training with biofeedback device — Use of the Smartphone application to perform a strengthening program for pelvic floor musculature, while using an intracavitary biofeedback device that will inform about vaginal pressure.
  Arms: Experimental group 1
Behavioral: Pelvic floor muscle training — Use of the Smartphone application to perform a strengthening program for pelvic floor musculature.
  Arms: Experimental group 2
Behavioral: Information about pelvic floor and communication with health professionals — Use of the Smartphone application with access to information about pelvic floor and direct communication with healthcare team.

SUMMARY:
Pelvic floor dysfunctions (PFD) are especially prevalent among females. As conservative management, strengthening pelvic floor (PF) musculature under health supervision, regard an important research line. However, embarrassment of female athletes limits healthcare demands. New technologies could facilitate an autonomous but supervised tele-rehabilitation programs.

This study will evaluate the effects of a 6-weeks strengthening PF program by using tele-rehabilitation, with or without intracavitary biofeedback, in the PF anatomo-functional characteristics, quality of life and sports performance of female athletes with PFD.

To this end, 45 female athletes with self-reported PFD who train and compete in athletic in Spain will be recruited and randomly distributed in three groups of the experimental study. During 6 weeks, all participants will use an specifically developed Smartphone application (named ACTITUD): the control group (CG) will have access to information about PF and direct communication with healthcare team; experimental group 1 (EG1) will have access to the same information and communication, and will perform a strengthening program for PF, which will be instructed by 3D avatars, while using an intracavitary biofeedback device that will inform about vaginal pressure; the experimental group 2 (EG2) will be similar to EG1, but they will not use the intracavitary biofeedback device.

Before and after these 6 weeks, anatomo-functional PF characteristics, quality of life, PFD symptoms and sports performance of all participants will be evaluated. As an additional outcome, the level of engagement of the athletes from experimental groups to complete the training program will be registered.

DETAILED DESCRIPTION:
Female athletes from EG1 and EG2 will complete the strengthening program for PF three times per week, during six weeks. Each session will last about 20 minutes and exercises will be modified every two weeks to meet the principle of training progression and avoid athletes become bored.

ELIGIBILITY:
Inclusion Criteria:

* To train and compete in any of the Track and Field modalities
* To have sports license from regional or national Track and Field Federation in the season when study starts.
* To have a self-reported pelvic floor disorder (urinary incontinence, fecal incontinence, sexual dysfunction or pelvic organ prolapse).

Exclusion Criteria:

* To have pelvic pain during the last three months.
* To have recurrent infections of urinary tract during the last three months.
* To be receiving physiotherapy treatment due to any pelvic floor disorder at the moment of the start of the study.
* To have been pregnant during the year prior to the start of the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Functional characteristics of pelvic floor musculature with perineometer | 6 weeks
  Change in the maximal voluntary contraction (MVC) according to the values of pressure collected by a perineometer (in mmHg) after the intervention period and compared to the athletes from the rest of groups. To assess it, participants will perform a maximal contraction of pelvic floor musculature during 3 seconds (three trials with 60 seconds apart). The best trial (the highest pressure) will be collected, as well as the rest vaginal pressure before the first trial of MVC.
Anatomical characteristics of pelvic floor structures with ultrasound I | 6 weeks
  Change in the levator hiatus length (in mm) after the intervention period and compared to the athletes from the rest of groups. This variable will be assessed by using transperineal approach with transducer in longitudinal orientation, at three different functional situations: at rest, while participants perform a maximal voluntary contraction (MVC) of the pelvic floor musculature, and also at straining.
Anatomical characteristics of pelvic floor structures with ultrasound II | 6 weeks
  Change in the anorectal angle (in degrees) and pubourethral angle (in degrees) after the intervention period and compared to the athletes from the rest of groups. These variables will be assessed by using transperineal approach with transducer in longitudinal orientation, at three different functional situations: at rest, while participants perform a maximal voluntary contraction (MVC) of the pelvic floor musculature, and also at straining.
Anatomical characteristics of pelvic floor structures with ultrasound III | 6 weeks
  Change in the symmetry of the bladder base (in mm) at rest and bladder base displacement (in mm) while participants perform a MVC of the pelvic floor musculature (PFM) and also during straining, after the intervention period and compared to the athletes from the rest of groups. These variables will be assessed by using a transabdominal approach with transducer, in transverse orientation.
Sports performance through maximal vertical jump | 6 weeks
  Change in the maximal height that athletes reach with a vertical jump (in meters) after the intervention period and compared to the athletes from the rest of groups. To assess it, participants will perform a maximal countermovement jump (three trials with 30 seconds apart). It will be collected the average of the three trials.
Presence of pelvic floor disorders symptomatology | 6 weeks
  Change in self-reported PFD symptoms through the PFD-SENTINEL questionnaire, after the intervention period and compared to the athletes from the rest of groups. To this end, athletes will reply the proposed PFD-SENTINEL tool consisting of 5 symptoms (urinary incontinence, anal incontinence, pelvic pain, pelvic organ prolapse, and overactive bladder syndrome) and 28 items. The responses to each item are categorized in yes or no. One point will be assigned for the affirmative response to each item. It will be considered the symptom score (presence or not of PFD symptoms),and total score (from 0 to 28 points).
Frequency of pelvic floor disorders symptomatology | 6 weeks
  In case of affirmative response to the presence of one or more PFD symptoms, it will be explore the frequency of the existing symptom. The responses will be graded on a 4-point scale indicating how often women have each symptom (1 = rarely, 2 = sometimes, 3 = often, and 4 = always). It will be explored the change after the intervention period and compared to the athletes from the rest of groups.
Sexual dysfunction symptomatology | 6 weeks
  Change in self-reported sexual dysfunction symptoms through The Female Sexual Function Index (FSFI), after the intervention period and compared to the athletes from the rest of groups. This scale consists of 19 items that assess sexual function over the past 4 weeks and yield domain scores in six areas: sexual desire, arousal, lubrication, orgasm, satisfaction, and pain. The responses to each item are graded as follows: 1 = never or very low, 2 = rarely or low, 3 = sometimes or moderate, 4 = often or high, 5 = always or very high. It will be consider individual score for each area (max 6 points) and total score (max 36 points).
Level of quality of life | 6 weeks
  It will be explore the change in quality of life due to the pelvic floor disorders symptoms (according to a scale from 0, no affection, to 10, maximal affection) after the intervention period and compared to the athletes from the rest of groups.

SECONDARY OUTCOMES:
Engagement to training program | 6 weeks
  Percentage of training program sessions that athletes from experimental groups completed during the six weeks of intervention, according to the number of proposed sessions (three times per week).

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Romero-Franco, Principal Investigator — University of the Balearic Islands
Locations (1):
- University of the Balearic Islands, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rodriguez-Lopez ES, Acevedo-Gomez MB, Romero-Franco N, Basas-Garcia A, Ramirez-Parenteau C, Calvo-Moreno SO, Fernandez-Dominguez JC. Urinary Incontinence Among Elite Track and Field Athletes According to Their Event Specialization: A Cross-Sectional Study. Sports Med Open. 2022 Jun 15;8(1):78. doi: 10.1186/s40798-022-00468-1. PMID 35704136
- [Result] Romero-Franco N, Molina-Mula J, Bosch-Donate E, Casado A. Therapeutic exercise to improve pelvic floor muscle function in a female sporting population: a systematic review and meta-analysis. Physiotherapy. 2021 Dec;113:44-52. doi: 10.1016/j.physio.2021.04.006. Epub 2021 Apr 29. PMID 34555673